CLINICAL TRIAL: NCT06724536
Title: Interaction Between Gut Microbiota and Tyrosine Kinase Inhibitors in Defining the Clinical Outcomes of Patients With Chronic Myeloid Leukemia
Brief Title: Interaction Between Gut Microbiota and TKIs in Defining the Clinical Outcomes of Patients With CML
Acronym: MICROBIO-LMC
Status: Recruiting | Type: Observational
Sponsor: Carmen Fava (Other)
Collaborators: Pfizer (Industry); Novartis (Industry)
Responsible Party: Sponsor-Investigator, Carmen Fava, Professor, University of Turin, Italy
Organization: University of Turin, Italy (Other)
Other Study IDs: MICROBIO-LMC
Record Dates: First submitted 2024-12-04; First posted 2024-12-09 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Leukemia,Myeloid, Chronic
Keywords: chronic myeloid leukemia; gut; microbiota; tyrosine kinase inhibitors
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, plasma and feces
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: non interventional study with the use of biological samples. — Patients will undergo to the follow evaluations:
  Gut microbiome on stool samples by NGS (16S rRNA gene amplicon sequencing); Markers of impaired intestinal permeability [diaminoxidase (DAO), serum zonulin], and markers of inflammation of the GI tract (fecal calprotectin); Plasma inflammatory indices, cytokines (by Luminex), markers of autoimmunity, and metabolic profile; Acquired and adaptive immunity by multiparametric flow cytometry on PB samples.

SUMMARY:
Gut microbiome (GM) is acquiring increasing importance in human health and disease. GM influences hematopoiesis and immune cells types differentiation. Patients with cancer are characterized by dysbiosis and compromised immunity. In the case of Chronic Myeloid Leukemia (CML), treatment with Tyrosine Kinase Inhibitors (TKIs) restores immunosurveillance; in particular deep molecular response (DMR) is associated with increased levels of NK and CD8+ Tcells. There is no literature on the effects of GM on CML outcomes. This project aims to identify a microbial signature associated with a higher probability of achieving DMR.

DETAILED DESCRIPTION:
Philadelphia positive Chronic Myeloid Leukemia (CML) is a myeloproliferative disorder originating from pluripotent hematopoietic cells. Treatment typically involves tyrosine-kinase inhibitors (TKIs), which have significantly improved long-term survival. While generally well-tolerated, TKIs can cause side effects, particularly gastrointestinal issues (diarrhea, constipation, abdominal pain, malabsorption, bleeding) and liver/pancreatic enzyme increases, which may persist and affect quality of life. Additionally, cardiovascular events, often linked to metabolic changes (e.g., glucose intolerance, diabetes, hypertension), occur more frequently during treatment. These side effects raise concerns about TKIs potentially inducing a chronic inflammatory response.

Recent research on the human microbiota highlights its importance in health. The microbiota plays a critical role in gut health, immune function, and metabolic processes, and its imbalances (dysbiosis) can contribute to a range of diseases. Factors such as diet, age, physical activity, and medication use can disrupt the microbiota. However, the relationship between gut microbiota and TKIs in CML patients remains unexplored.

The current study will evaluate by whether different CML gut microbiota genotypes influence TKI treatment responses, whether microbiota alterations cause inflammation or metabolic disorders, and whether microbiota, along with dysmetabolism and dysimmunity, contribute to variations in treatment efficacy and tolerance

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old
* Chronic Myeloid Leukemia Patients
* Any stage of the disease

Exclusioni Criteria:

none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All hematologic patients of the the Hematology Division of the AO Ordine Mauriziano di Torino with a diagnosis of Philadelphia positive Chronic Myeloid Leukemia (CML) will be included.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
genotypes of the intestinal microbiota and responses to treatment with TKI. | 4 years
  The primary objective is to assess the association between genotypes of the intestinal microbiota (in eubiosis or dysbiosis) of patients with CML and responses (efficacy and tolerability in the short and long term) to treatment with TKI.

CONTACTS AND LOCATIONS:
Overall Officials: Carmen Fava, Principal Investigator — Department of Clinical and Biological Sciences, University of Turin, Turin, Italy
Locations (1):
- AO Ordine Mauriziano di Torino, Torino, Italy

IPD SHARING:
Plan to Share IPD: No